CLINICAL TRIAL: NCT00765206
Title: Randomized, Crossover Pharmacodynamic Study Comparing the Effects of Zegerid® (20 mg Omeprazole/Sodium Bicarbonate) and Prilosec OTC® Tablets (20 Mg-equivalent Omeprazole)
Brief Title: A Pharmacodynamic Study Comparing Zegerid® and Prilosec OTC® (Study CL2008-02)(P07814)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 18134; CL2008-02; P07814 (Other: Merck)
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Acid; Human Experimentation
MeSH Terms: interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zegerid (Experimental): Omeprazole 20 mg /sodium bicarbonate 1100 mg over-the-counter (OTC) Capsule
  Interventions: Drug: Omeprazole/sodium bicarbonate
- Prilosec (Active Comparator): Omeprazole magnesium 20 mg OTC tablet
  Interventions: Drug: omeprazole magnesium (20 mg equivalent)

INTERVENTIONS:
Drug: Omeprazole/sodium bicarbonate — Single dose of omeprazole/sodium bicarbonate per day for either 1 or 7 days.
  Other Names: Zegerid
  Arms: Zegerid
Drug: omeprazole magnesium (20 mg equivalent) — Single dose of omeprazole magnesium per day for either 1 or 7 days.
  Other Names: Prilosec OTC Tablet
  Arms: Prilosec

SUMMARY:
Open-label randomized crossover design study. 60 participants will be evaluated on Day 1 to compare effects on stomach acid; 30 participants will continue treatment for 7 days and will have repeat evaluations at Day 7.

DETAILED DESCRIPTION:
Enrolled participants were divided into 2 groups, with 30 participants in each group.

Group 1: This group was randomized into a single-dose, 2-way crossover design. These participants received single administrations (day 1 dosing only) of Zegerid OTC Capsules, and Prilosec OTC Tablets (both at a 20 mg omeprazole dose), in a 2-way randomized order, with a minimum of a 2-week washout period between treatment legs. This group underwent a 24-hour intragastric pH study on each of the 2 dosing occasions.

Group 2: This group was randomized into a 2-way crossover design in which they received 7 days administration of Zegerid OTC Capsules and Prilosec OTC Tablets, respectively. As with the prior group, there was a minimum of a 2-week washout period between treatment legs. Participants assigned to this treatment group underwent 24-hour intragastric pH recordings on the days which they received their 1st and last (7th) dose of the two treatment drugs.

In addition to the above detailed procedures, all participants (both groups) underwent a 24-hour baseline intragastric pH study prior to starting their randomized treatments. This study design enabled all 60 participants to be evaluated for effects of the first dose of Prilosec OTC Tablets and Zegerid OTC Capsules on change in intragastric pH during the subsequent 24-hour period following the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects who are 18-65 years of age.
* Non-childbearing potential females or those using birth control.

Exclusion Criteria:

* History of hypersensitivity, allergy or intolerance to omeprazole or other proton pump inhibitors
* History of significant gastrointestinal disease
* Any significant medical illness
* Gastrointestinal disorder or surgery leading to impaired drug absorption
* Currently using gastrointestinal medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were enrolled: 30 participants were randomized to 1-Day Dosing and 30 participants were randomized to 7-Day Dosing. This was a crossover study, ie, participants in both groups received one treatment [Zegerid or Prilosec], followed by a 2-week washout period, followed by the other treatment [Prilosec or Zegerid].
Groups:
- Zegerid First, Then Prilosec (1- Day Dosing): Participants received Zegerid Over-the-counter (OTC) Capsules (omeprazole 20 mg and sodium bicarbonate 1100 mg) in the first intervention and Prilosec OTC Tablets (omeprazole 20 mg) in the second intervention (after washout period)
- Prilosec First, Then Zegerid (1-Day Dosing); Prilosec First, Then Zegerid (7-Day Dosing): Participants received Prilosec OTC Tablets (omeprazole 20 mg) in the first intervention and Zegerid OTC Capsules (omeprazole 20 mg and sodium bicarbonate 1100 mg) in the second intervention (after washout period)
- Zegerid First, Then Prilosec ( 7-Day Dosing): Participants received Zegerid OTC Capsules (omeprazole 20 mg and sodium bicarbonate 1100 mg) in the first intervention and Prilosec OTC Tablets (omeprazole 20 mg) in the second intervention (after washout period)
Period: First Intervention
Arm/Group | Zegerid First, Then Prilosec (1- Day Dosing) | Prilosec First, Then Zegerid (1-Day Dosing) | Zegerid First, Then Prilosec ( 7-Day Dosing) | Prilosec First, Then Zegerid (7-Day Dosing)
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 14 Days
Arm/Group | Zegerid First, Then Prilosec (1- Day Dosing) | Prilosec First, Then Zegerid (1-Day Dosing) | Zegerid First, Then Prilosec ( 7-Day Dosing) | Prilosec First, Then Zegerid (7-Day Dosing)
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Zegerid First, Then Prilosec (1- Day Dosing) | Prilosec First, Then Zegerid (1-Day Dosing) | Zegerid First, Then Prilosec ( 7-Day Dosing) | Prilosec First, Then Zegerid (7-Day Dosing)
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Median 24-hour Intragastric pH on the 7th Day of Drug Administration
Description: The change from Baseline in median pH was calculated as: median pH on Day 7 minus median pH at Baseline. The pH scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic. A pH greater than 7 is basic.
Time Frame: Baseline and 7 days
Measure: Median (Full Range); unit: pH scale
Groups:
- Zegerid: Participants in the 7-Day Dosing group. Measurements taken on the 7th day of Zegerid administration.
- Prilosec: Participants in the 7-Day Dosing group. Measurements taken on the 7th day of Prilosec administration.
Arm/Group | Zegerid | Prilosec
Number analyzed (Participants) | 30 | 30
pH scale
  Day 7 Score | 4.575 (1.349) [1.33 to 5.98] | 3.980 (1.433) [1.37 to 5.94]
  Change from Baseline in pH | 3.165 (1.360) [0.03 to 4.75] | 2.550 (1.478) [-0.89 to 4.46]

ADVERSE EVENTS:
Groups:
- Zegerid: Subjects who received a single dose of Zegerid per day for either 1 or 7 days.
- Prilosec: Subjects who received a single dose of Prilosec per day for either 1 or 7 days.
Arm/Group | Zegerid | Prilosec
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Schering-Plough HealthCare Products, Inc. reserves all publication and

presentation rights.